CLINICAL TRIAL: NCT02557698
Title: Prospective, Randomized Study on the Skin Functional Parameters to Assess Skin Barrier Improvement After the Use of a Commercially Available Oil Bath Containing 84.75% Soybean Oil Compared to no Bath Additive
Brief Title: Effectiveness of Using an Oil Bath Additive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, PD Dr. Jan Kottner, Scientific Director Clinical Research Center for Hair and Skin Science, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC-SP-ABC-13
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Xerosis Cutis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balneum oil bath (Experimental): Balneum oil bath, bathing every other day for four weeks
  Interventions: Other: Balneum oil bath
- standard skin cleanser (No Intervention): Usual skin cleanser (non-oil containing), bathing or showering every other day for four weeks

INTERVENTIONS:
Other: Balneum oil bath
  Arms: Balneum oil bath

SUMMARY:
Epidermis that lacks moisture and/or sebum presents as dry skin, which is often characterized by a pattern of fine lines, scaling and itching. In dry skin, the barrier function may be compromised. Skin care practices to decrease the risk of development of dry skin and/or to improve dry skin condition have barely been investigated. Bathing with bath oils has been shown to increase skin hydration, thus helping to stabilize skin barrier function. Therefore, the aim of this study is to investigate the effect of bathing every other day on the skin barrier. Functional parameters, such as TEWL, stratum corneum hydration (SCH) and skin-pH (pH) were measured to characterize skin barrier function.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, or children whose parent(s) or guardian(s) have given their written informed consent for their child's participation in the study
* Child specific written informed consent, if over 7 years of age
* Subjects with a general good and stable health condition
* Subjects with clinically stable medical conditions
* Accept to abstain from sunbathing and solarium during the study
* Overall Dry Skin score (ODS) of 1 to 2 at arms and lower legs
* TEWL > 12 g/m2/h on the left mid volar forearm

Exclusion Criteria:

* Any dermatological condition or skin affection which may interfere with the study assessments, e.g. scars
* Suffering from porphyria
* Suffering from severe photodermatoses according to the judgment of the investigator
* Clinically significant, possibly unstable medical conditions such as metastatic tumor
* Currently having other malignant or benign tumors of the skin in the investigational area
* Any other acute or chronic pathology that may interfere with the study conduct in the investigator's opinion
* Known allergy or intolerance to any ingredients of the study product, e.g. propylene glycol
* Use of (medical) oil-containing bath additives or other oil-containing cleansers
* Current topical or systemic treatment affecting the skin, e.g. diuretics
* Treatment of dry and/or inflammatory skin conditions with topical corticosteroids during the 4 weeks before inclusion
* Systemic immunosuppressive or immunomodulatory therapy
* Topical retinoids applied during the 6 weeks before inclusion
* Topical application of immunosuppressive treatment during the 6 weeks before inclusion
* Therapeutic UV-Radiation during the 6 weeks before inclusion
* Increased UV-exposure during the 6 weeks before inclusion

Ages: 6 Months to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Kottner J, Kanti V, Dobos G, Hahnel E, Lichterfeld-Kottner A, Richter C, Hillmann K, Vogt A, Blume-Peytavi U. The effectiveness of using a bath oil to reduce signs of dry skin: A randomized controlled pragmatic study. Int J Nurs Stud. 2017 Jan;65:17-24. doi: 10.1016/j.ijnurstu.2016.10.010. Epub 2016 Oct 26. PMID 27815985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitmant period: Nov 2014 - Apr 2015, Location: Charité University Hospital
Groups:
- Balneum Oil Bath: Balneum oil bath, bathing every other day for four weeks
  Balneum oil bath
Period: Overall Study
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.0 [13.3 to 70.0] | 29.5 [6.0 to 68.3] | 32.5 [8.3 to 69.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intervention group: 30 control group: 30
  Participants
    Female | 12 | 15 | 27
    Male | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h at the Left Mid Volar Forearm
Description: TEWL was measured using the Tewameter TM300 (Courage+Khazaka, Cologne, Germany) according to international guidelines (Rogiers 2001). This open chamber intrument measured water evaporation from the skin by temperature and humidity sensors inside the cylinder. Means of triple measurements per skin area in g/m2/h on the left midvolar forearm.
  Visit 3 (day 28) - end of study visit
Time Frame: Day 28 +/- 3
Population: Male or female gender, aged between 6 months and 85 years
Measure: Mean (Standard Deviation); unit: g/m2/h
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
g/m2/h | 10.0 (2.0) | 11.9 (2.5)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; H0=Intervention and control groups do not differ with respect to the TEWL forearm at visit 3 H1=The TEWL on the forearm at visit 3 differs between the groups; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.1 to -0.8]

2. Secondary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h at the Left Mid Volar Forearm
Description: TEWL was measured using the Tewameter TM300 (Courage+Khazaka, Cologne, Germany) according to international guidelines (Rogiers 2001). This open chamber intrument measured water evaporation from the skin by temperature and humidity sensors inside the cylinder. Means of triple measurements per skin area in g/m2/h on the left midvolar forearm.
  Visit 2 (day14) - intermediate visit
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: g/m2/h
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
g/m2/h | 9.7 (2.2) | 12.0 (2.3)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-3.5 to -1.2]

3. Secondary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h at the Right Lateral Lower Leg
Description: TEWL was measured using the Tewameter TM300 (Courage+Khazaka, Cologne, Germany) according to international guidelines (Rogiers 2001). This open chamber intrument measured water evaporation from the skin by temperature and humidity sensors inside the cylinder. Means of triple measurements per skin area in g/m2/h at the right lateral lower leg.
  Visit 2 (day14)
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: g/m2/h
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
g/m2/h | 9.0 (1.9) | 10.7 (3.6)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.024, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.2 to -0.2]

4. Secondary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h at the Right Lateral Lower Leg
Description: TEWL was measured using the Tewameter TM300 (Courage+Khazaka, Cologne, Germany) according to international guidelines (Rogiers 2001). This open chamber intrument measured water evaporation from the skin by temperature and humidity sensors inside the cylinder. Means of triple measurements per skin area in g/m2/h at the right lateral lower leg.
  Visit 3 (day 28)
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: g/m2/h
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
g/m2/h | 9.3 (2) | 11.0 (3.2)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.1 to -0.3]

5. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Right Lateral Lower Leg
Description: SCH was measured using the Corneometer (Courage+Khazaka, Cologne, Germany) according to international guidelines which measured the hydratation level of the stratum corneum as electrical capacitance (Berardesca et al. 1997). The higher the values, the higher the SCH. Per investigational site three replicate measurements were carried out.
  Visit 2 (day 14)
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Arbitrary Units | 29.9 (6.7) | 30.0 (8)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.964, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-3.9 to 3.7]

6. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Right Lateral Lower Leg
Description: SCH was measured using the Corneometer (Courage+Khazaka, Cologne, Germany) according to international guidelines which measured the hydratation level of the stratum corneum as electrical capacitance (Berardesca et al. 1997). The higher the values, the higher is SCH. Per investigational site three replicate measurements were carried out.
  Visit 3 (day 28)
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Arbitrary Units | 32.3 (7.7) | 28.0 (7.1)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.025, t-test, 2 sided; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [0.5 to 8.2]

7. Secondary Outcome: Skin Surface Mean Roughness (Ra) in µm at the Right Lateral Lower Leg
Description: Skin roughness was measured using the Visioscan VC98 (Courage+Khazaka, Cologne, Germany). It consists of a UV light camera and measures the skin surface profiles. Ra=mean roughness
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 16.7 (2.9) | 17.3 (4.0)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.458, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.5 to 1.1]

8. Secondary Outcome: Skin Surface Mean Roughness (Ra) in µm at the Right Lateral Lower Leg
Description: as for outcome 7
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 16.7 (2.9) | 18.4 (4.1)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.066, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.5 to 0.1]

9. Secondary Outcome: Skin Surface Mean Roughness (Rz) in µm at the Right Lateral Lower Leg
Description: Skin roughness was measured using the Visioscan VC98 (Courage+Khazaka, Cologne, Germany) device. It consists of a UV light camera and measures the skin surface profiles. The parameter Rz was calculated. Rz=mean roughness of five equally spaced sampling lenghts.
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 70.1 (11.6) | 75.1 (18.9)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.171, t-test, 2 sided; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-13.7 to 2.5]

10. Secondary Outcome: Skin Surface Mean Roughness (Rz) in µm at the Right Lateral Lower Leg
Description: as for outcome 9
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 72.1 (13.0) | 79.6 (16.9)
Statistical Analysis 1: Comparison: Balneum Oil Bath; Test type: Superiority or Other; p = 0.059, t-test, 2 sided; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-15.3 to 0.3]

11. Secondary Outcome: Skin Surface pH at the Right Lateral Lower Leg
Description: Skin surface pH was measured using the Skin-pH-Meter PH905 (Courage+Khazaka, Cologne, Germany) according to international guidelines (Parra et al. 2003). The pH of the skin surface may differ from the pH of the stratum corneum. Means of triple measurements/images per skin area.
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: non-dimensional
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
non-dimensional | 5.4 (0.7) | 5.3 (0.5)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.400, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.5]

12. Secondary Outcome: Skin Surface pH at the Right Lateral Lower Leg
Description: as for outcome 11
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: non-dimensional
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
non-dimensional | 5.2 (0.5) | 5.1 (0.4)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.100, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.4]

13. Secondary Outcome: Overall Dry Skin (ODS) Score at the Left Arm
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks) Visit 2 (day14) - intermediate visit
Time Frame: Day 14 +/- 2
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 7 | 7
  ODS score 1 | 19 | 19
  ODS score 2 | 4 | 4
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Overall Dry Skin (ODS) Score at the Left Arm
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness by the investigator using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks)
Time Frame: Day 28 +/- 3
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 13 | 13
  ODS score 1 | 14 | 13
  ODS score 2 | 3 | 4
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.914, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Overall Dry Skin (ODS) Score at the Right Arm
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks) Visit 2 (day14)
Time Frame: Day 14 +/- 2
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 8 | 6
  ODS score 1 | 18 | 20
  ODS score 2 | 4 | 4
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.822, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Overall Dry Skin (ODS) Score at the Right Arm
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks) Visit 3 (day 28)
Time Frame: Day 28 +/- 3
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 12 | 9
  ODS score 1 | 14 | 18
  ODS score 2 | 4 | 3
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.585, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Overall Dry Skin (ODS) Score at the Left Lower Leg
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks) Visit 2 (day 14) - intermediate visit
Time Frame: Day 14 +/- 2
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 4 | 2
  ODS score 1 | 17 | 13
  ODS score 2 | 9 | 15
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.259, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Overall Dry Skin (ODS) Score at the Left Lower Leg
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks) Visit 3 (day 28) - end of study visit
Time Frame: Day 28 +/- 3
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 2 | 4
  ODS score 1 | 17 | 14
  ODS score 2 | 11 | 11
  ODS score 3 | 0 | 1
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.581, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Overall Dry Skin (ODS) Score at the Right Lower Leg
Description: as for outcome 17
Time Frame: Day 14 +/- 2
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 4 | 2
  ODS score 1 | 16 | 11
  ODS score 2 | 10 | 17
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.182, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Overall Dry Skin (ODS) Score at the Right Lower Leg
Description: as for outcome 16
Time Frame: Day 28 +/- 3
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 3 | 3
  ODS score 1 | 16 | 14
  ODS score 2 | 11 | 12
  ODS score 3 | 0 | 1
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.759, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Overall Dry Skin (ODS) Score at the Trunk
Description: The Overall Dry Skin score is a standardized instrument to clinically assess the presence or severity of skin dryness using a five point rating scale according to Serup1995, Kang et al. 2014 on both arms, lower legs and trunk.
  (0=Absent, 1=Faint scaling, faint roughness and dull appearance, 2=Small scales in combination with a few larger scales, slight roughness and whitish appearance, 3=Small and larger scales uniformly distributed, definite roughness, possibly slight redness and possibly a few superficial cracks, 4=Dominated by large scales, advanced roughness, redness present, eczematous changes and cracks) Visit 2 (day 14)
Time Frame: Day 14 +/- 2
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Participants
  ODS score 0 | 13 | 14
  ODS score 1 | 15 | 15
  ODS score 2 | 2 | 1
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.831, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Overall Dry Skin (ODS) Score at the Trunk
Description: as for outcome 18
Time Frame: Day 28 +/- 3
Population: ODS score 0-4
Measure: Count of Participants; unit: Participants
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 29 | 30
Participants
  ODS score 0 | 19 | 12
  ODS score 1 | 10 | 16
  ODS score 2 | 0 | 2
  ODS score 3 | 0 | 0
  ODS score 4 | 0 | 0
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.084, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Left Midvolar Forearm
Description: as for outcome 5
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Arbitrary Units | 37.3 (6.0) | 33.8 (8.7)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.07, t-test, 2 sided; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-0.3 to 7.4]

24. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Left Midvolar Forearm
Description: SCH was measured using the Corneometer (Courage+Khazaka, Cologne, Germany) according to international guidelines which measured the hydratation level of the stratum corneum as electrical capacitance (Berardesca et al. 1997). The higher the values, the higher the SCH. Per investigational site three replicate measurements were carried out.
  Visit 3 (day 28)
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
Arbitrary Units | 38.2 (7.4) | 34.1 (6.7)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.029, t-test, 2 sided; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [0.4 to 7.7]

25. Secondary Outcome: Skin Surface Mean Roughness (Ra) in µm at the Left Midvolar Forearm
Description: as for outcome 7
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 16.5 (2.6) | 17.1 (2.1)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.325, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.8 to 0.6]

26. Secondary Outcome: Skin Surface Mean Roughness (Ra) in µm at the Left Midvolar Forearm
Description: as for outcome 7
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 17.4 (4.0) | 18.2 (3.0)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.365, t-test, 2 sided; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.6 to 0.9]

27. Secondary Outcome: Skin Surface Mean Roughness (Rz) in µm at the Left Midvolar Forearm
Description: as for outcome 9
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 66.7 (8.3) | 70.4 (10.6)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.143, t-test, 2 sided; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-8.5 to 1.3]

28. Secondary Outcome: Skin Surface Mean Roughness (Rz) in µm at the Left Midvolar Forearm
Description: as for outcome 9
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
µm | 69.7 (12.2) | 70.9 (8.1)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.662, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-6.5 to 4.2]

29. Secondary Outcome: Skin Surface pH at the Left Midvolar Forearm
Description: Skin surface pH was measured using the Skin-pH-Meter PH905 (Courage+Khazaka, Cologne, Germany) according to international guidelines (Parra et al. 2003). The pH on the skin surface may differ from the pH of the stratum corneum. Means of triple measurements/images per skin area.
Time Frame: Day 14 +/- 2
Measure: Mean (Standard Deviation); unit: non-dimensional
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
non-dimensional | 5.1 (0.6) | 5.3 (0.5)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.326, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1]

30. Secondary Outcome: Skin Surface pH at the Left Midvolar Forearm
Description: as for outcome 29
Time Frame: Day 28 +/- 3
Measure: Mean (Standard Deviation); unit: non-dimensional
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Number analyzed (Participants) | 30 | 30
non-dimensional | 5.2 (0.6) | 5.1 (0.5)
Statistical Analysis 1: Comparison: Balneum Oil Bath vs Standard Skin Cleanser; Test type: Superiority or Other; p = 0.687, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.4]

ADVERSE EVENTS:
Arm/Group | Balneum Oil Bath | Standard Skin Cleanser
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No